CLINICAL TRIAL: NCT06669767
Title: Behavioral Indicators of Pain Representation
Acronym: ICOR
Status: Completed | Type: Observational
Sponsor: Universite de Picardie Jules Verne (Other)
Responsible Party: Principal Investigator, Adrien Hakimi, Research engineer, Universite de Picardie Jules Verne
Other Study IDs: IRB00012476_2024_10_07_328
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Non-specific Chronic Low Back Pain; Healthy Volunteer
Keywords: Kinesiophobia; Low back pain; Posturography
MeSH Terms: conditions — Kinesiophobia; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-specific chronic low back pain: Participants with non-specific chronic low back pain (>3 months).
- Control group: Healthy volunteers, without any low back pain.

SUMMARY:
The goal of this observational study is to compare the postural response to the mental simulation of everyday situations identified as painful in participants with non-specific low back pain and healthy volunteers.

The main questions it aims to answer are :

Do participants with low-back pain show reduced variability in center of pressure displacements compared with non-painful participants when faced with mental simulation of everyday situations identified as painful? Is the postural response correlated with the level of kinesiophobia? Participants will be faced to pictures of everyday situations identified as painful while several physiological measurements (posturography, electromyography, heart rate) are being recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55
* Non-specific chronic low back pain for the concerned group

Exclusion Criteria:

* Low back pain for 0 to 3 months
* Unable to stand 1 minute without technical aid
* Neurological, motor or cognitive know impairment
* BMI > 30

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male/Female
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Standard deviation of the position of the center of pressure on the anteroposterior axis (SD-COP-AP) | Baseline
  Movements of the center of pressure (COP) are recorded using a force plate, and the SD-COP-AP is calculated after recording and is an indicator of the postural response.

SECONDARY OUTCOMES:
Mean position of the center of pressure on the anteroposterior axis (COP-AP) | Baseline
Mean position of the center of pressure on the mediolateral axis (COP-ML) | Baseline
Standard deviation of the position of the center of pressure on the mediolateral axis (SD-COP-ML) | Baseline
Sway length of the center of pressure on the anteroposterior axis (L-COP-AP) | Baseline
Sway length of the center of pressure on the mediolateral axis (L-COP-ML) | Baseline
Tibialis anterior muscle activity | Baseline
  Measured by electromyography, RMS normalized to maximum voluntary contraction.
Soleus muscle activity | Baseline
  Measured by electromyography, RMS normalized to maximum voluntary contraction.
Longissimus dorsi muscle activity | Baseline
  Measured by electromyography, RMS normalized to maximum voluntary contraction.
Co-activation (Soleus/Tibialis anterior) | Baseline
Coefficient of variation for muscle activity of tibialis anterior | Baseline
Coefficient of variation for muscle activity of soleus | Baseline
Coefficient of variation for muscle activity of longissimus dorsi | Baseline
Mean heart rate | Baseline
Mean RR interval | Baseline
Standard deviation of normal RR intervals (SDNN) | Baseline
Root mean square of successive R-R intervals (RMSSD) | Baseline
Power of very low frequency from frequency analysis (VLF) | Baseline
Power of low frequency from frequency analysis (LF) | Baseline
Power of high frequency from frequency analysis (HF) | Baseline
Ratio of LF/HF (post-frequency analysis) | Baseline
Tampa scale for kinesiophobia (TSK) score | Baseline
  Kinesiophobia was evaluated with the Tampa Scale for Kinesiophobia (TSK), a self-administered questionnaire validated in French. The TSK measures the fear of movement and is used in various painful conditions. It includes 17 items evaluated on a 4-point Likert scale. The total score range is 17-68 and a high score indicates a greater fear of movement.
Brief pain inventory (BPI) score | Baseline
  Pain was assessed with the Brief Pain Inventory (BPI), a reliable self-administered questionnaire about pain severity (4 items) and interference with daily living (7 items) validated in French. Each item is evaluated on a numerical scale from 0 to 10. A high score indicates significant pain or significant interference in daily living.
EQ-5D-5L questionnaire score | Baseline
  The EQ-5D-5L is a standardized questionnaire used as a measure of health-related quality of life. The first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression, on a five-level scale (no problem, slight problems, moderate problems, severe problems, unable to). The second part consist in a visual analogic scale about global health of the participant and provide a value from 0 to 100 with high value representing a good health.
Fear-Avoidance Component Scale (FACS) score | Baseline
  The fear-avoidance component scale is used to measure the major fear-avoidance signs in painful conditions. It includes 20 items evaluated on a 5-point Likert scale. The total score is from 0 to 100 with 5 severity levels: 0-20 subclinical, 21-40 low, 41-60 moderate, 61-80 severe, and extreme 81-100.
Pain catastrophizing scale (PCS) score | Baseline
  Catastrophism was evaluated with the pain catastrophizing scale. It includes 13 items evaluated on a 4-point Likert scale and divided into 3 dimensions: magnification, rumination, and helplessness. A high score corresponds to a high level of catastrophism. The total score ranges from 0 to 52 with a cut-off score of 30 for a significant catastrophism level.
Hospital Anxiety and Depression scale (HAD) score | Baseline
  The Hospital Anxiety and Depression scale (HAD) includes 14 items, 7 for anxiety and 7 for depression validated in French. Each item is rated from 0 to 3 and the scores for each dimension range from 0 to 21. Cut-off scores were established with 8-10 being uncertain symptomatology and above 10 being definite symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LELARD, PhD, Study Director — Universite de Picardie Jules Verne
Locations (1):
- Université de Picardie Jules Verne, Amiens, France

IPD SHARING:
Plan to Share IPD: No